CLINICAL TRIAL: NCT04993300
Title: Repetitive Transcranial Magnetic Stimulation in Treatment of Taiwanese Amphetamine Users: A Pilot Study
Brief Title: Repetitive Transcranial Magnetic Stimulation in Amphetamine Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202010115DINA
Record Dates: First submitted 2021-07-21; First posted 2021-08-06 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Craving; Depression, Anxiety; Amphetamine Addiction
Keywords: Addiction; amphetamine; transcranial magnetic stimulation
MeSH Terms: conditions — Depression; Anxiety Disorders; Amphetamine-Related Disorders; Behavior, Addictive | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- transcranial magnetic stimulation (TMS) (Experimental): This arm constitute of methamphetamine users who undergone abstinent period
  Interventions: Device: transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Device: transcranial magnetic stimulation (TMS) — The methamphetamine user will undergo a one-month TMS intervention. In Week 1, subjects will attend continuously 5 daily TMS sessions. From Week 2 to Week 4, subjects are treated once a week. Each session will have 40 repeats of 4-second train and 15-sec train interval.

SUMMARY:
The study aims to test whether transcranial magnetic stimulation (TMS) improves the craving, depression, anxiety and cognitive function during the abstinent period of methamphetamine users.

DETAILED DESCRIPTION:
Background:

The disease burden of methamphetamine (MA) use is a critical issue in public health, while the abusers increased rapidly in recent years. The effect of medical intervention for MA addiction is still limited, and the cost of psychotherapy is high. In Taiwan, the MA defendant would be sent to the district inspection after the police confirmed the MA abuse. The prosecutor could assess the case to replace the penalty of imprisonment with a suspended sentence, which included one year of addiction treatment in the designated hospital. However, the insufficient treatment of MA addiction resulted in a subsequent high rescinded rate of suspended sentence cases and led people to doubt these medical intervention programs. Hence, the primary mission is to improve the treatment efficacy within the treatment program. Growing evidence has suggested the effectiveness of transcranial magnetic stimulation (TMS) in improving craving, affective symptoms, and cognitive impairment. However, the majority of the studies were conducted in China. Under China's legal system, researchers designed intense TMS treatment programs for MA users, which was not entirely applicable within Taiwan's system. Therefore, the current proposal aims to design a new TMS treatment and evaluate the tolerability, efficacy, and sustained effect of Taiwanese MA users within the suspended sentence.

Methods:

The investigators applied a case-only follow-up study and divided the study into two phases. Fifteen MA users within the suspended sentence who are under the outpatient-based MA abuse treatment program will be recruited. In Phase 1, 15 subjects will be randomly assigned to two TMS intensity groups (80% and 100%). After one TMS treatment session, subjects will be interviewed with the visual analog scale and the tolerability questionnaire to detect their side-effect and the primary effect of craving reduction. After evaluating the side-effect rate and the craving reduction effect, the investigators will select the subsequent TMS treatment program's intensity. In Phase 2, all subjects undergo a four-week TMS treatment program. In Week 1, subjects will attend continuously five daily TMS sessions. In Week 2 to Week 4, subjects are treated once a week. After 8 TMS sessions, the investigators will follow up one month and three months later. The investigators apply the Visual analog scale, Beck depression inventory, Beck anxiety inventory, and Continuous performance test in each intervention and follow-up time point to measure the efficacy and sustain effect of improving craving, depression, anxiety, and cognitive impairment.

ELIGIBILITY:
Inclusion criteria:

1. Age ranged 20-65.
2. Under judicially supervised outpatient-based methamphetamine abuse treatment program

Exclusion criteria:

1. Major disorders other than substance use disorders in Diagnostic and Statistics Manual-5 (e.g. Schizophrenia, organic brain syndrome, and bipolar disorders).
2. Epilepsy, head trauma, migraine, cardiovascular comorbidity, atypical parkinsonian disorder
3. patients with heart pacemakers, implanted drug delivery aids, artificial electronic ears, implantable defibrillators, and/or implanted nerve stimulators, and near the implants mentioned above.
4. patients who have metal implants in their bodies, as well as those with metal implants.
5. people who have damaged skin in areas of the patient's body that receive stimulation.
6. patients with multiple sclerosis.
7. patients who have extensive ischemic scarring.
8. pregnant women.
9. patients with a family history of spasms/epilepsy
10. patients taking medications that may lower the seizure threshold.
11. patients with severe sleep disorders related to previous rTMS treatment.
12. patients with severe heart disease
13. patients with intracranial stress caused by uncontrollable migraines.
14. people who have been evaluated by a physician as unfit to participate in clinical trials.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (Taiwanese version) | 20 weeks
  Respondents will specify their level of craving from none to extreme on a 100 mm line (score: 0-10) in each questionnaires, and there are nine questionnaires related to craving.

SECONDARY OUTCOMES:
The Beck depression inventory (Taiwanese version BDI) | 20 weeks
  The Beck depression inventory (Taiwanese version BDI) will be applied to evaluate the depression during the period of methamphetamine abstinence. (Total score: 0-63)
The Beck anxiety inventory (Taiwanese version BAI) | 20 weeks
  The Beck anxiety inventory (Taiwanese version BAI) will be applied to evaluate the anxiety during the period of methamphetamine abstinence. (Total score: 0-63)
Cognitive function | 20 weeks
  Continuous performance test was developed by Rosvold and designed as a computerized test of cognitive function.
Tolerance | 20 weeks
  The respondents will specify five physical symptoms which might related to rTMS intervention (Yes/No: headache, local pain/discomfort, head/face pain/discomfort, seizure, hearing loss/ear ache)

CONTACTS AND LOCATIONS:
Overall Officials: Chen Cheng-Che, MD,MSc, Principal Investigator — Physician, Department if Psychiatry, National Taiwan University Hospital - Biomedical Park Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan